CLINICAL TRIAL: NCT05975788
Title: Effect of Staphylococcus and Neisseria Tablets on Clinical Outcome Among Patients With Chronic Obstructive Pulmonary Disease: A Multi-center, Prospective Study
Brief Title: Effect of Staphylococcus and Neisseria Tablets on Clinical Outcome Among Patients With Chronic Obstructive Pulmonary Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Sun Yongchang, Director of Respiratory Department, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YL20230221
Record Dates: First submitted 2023-07-17; First posted 2023-08-04 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Staphylococcus and Neisseria group (Experimental): Experimental group will receive Staphylococcus and Neisseria Tablets (0.3mg/tablet) and standard care. Administration Staphylococcus and Neisseria is 4 tablets each time and 3 times a day, and treatment period ranges from 3 to 6 months.
  Interventions: Drug: Staphylococcus and Neisseria Tablets
- Standard care group (No Intervention): Standard care based on clinical experience without interventions.

INTERVENTIONS:
Drug: Staphylococcus and Neisseria Tablets — Staphylococcus and Neisseria tablets is used as an adjuvant treatment drug for respiratory disease in acute attack period, such as chronic tracheitis, bronchitis and various types of colds. It has been proved to effectively shorten the course of disease. In this study, Staphylococcus and Neisseria tablets will be administered with 4 tablets each time and 3 times a day, and treatment period ranges from 3 to 6 months according to clinicians.
  Arms: Staphylococcus and Neisseria group

SUMMARY:
This is a multi-center, prospective study. This study aims to investigate the incidence of acute exacerbation within 12 months, as well as the safety of Staphylococcus and Neisseria Tablets on patients with chronic obstructive pulmonary disease (COPD). In addition, this study investigates the improvement of hospitalization, improvement of pulmonary function, improvement of symptoms, and the use of anti-Infective drugs among COPD patients.

DETAILED DESCRIPTION:
A total of 750 eligible COPD patients were enrolled, and were randomly divided into experimental group and control group with a ratio of 2:1. Experimental group will receive Staphylococcus and Neisseria Tablets (0.3mg/tablet) and standard care. Drug administration is 4 tablets each time and 3 times a day, and treatment period ranges from 3 to 6 months. Control group will receive standard care without interventions.

All participants have to sign informed consent. After baseline (V0/V1), participants will be followed up for 12 months with four follow-up visits at 4 weeks ± 14d (V2), 13 weeks ± 14d (V3), 26 weeks ± 14d (V4), and 52 weeks ± 14d (V5). Among them, V2 can be phone interview.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years, males and females.
* Clinical diagnosis of COPD, defined as FEV1/FVC<70% after inhaling bronchodilators.
* At least 1 moderate to severe acute exacerbation of COPD in the past year.
* Patient or their legal agent sign informed consent with a date after understanding the purpose and procedures of the research, and be willing to participate in the study.

Exclusion Criteria:

* Patients with active pulmonary tuberculosis, asthma, or uncontrolled advanced malignant tumors; or after partial, lobar, or total pneumonectomy.
* Patients with acute cardio cerebral vascular disease such as acute myocardial infarction, acute stroke and acute heart failure.
* Patients with liver failure or renal failure and need blood purification treatment.
* Patients with rheumatic diseases and autoimmune diseases.
* Have participated or currently in interventional clinical trials within 30 days.
* Patients with previous (within 3 months before signing the informed consent) or current use of immunomodulatory drugs (including thymosin, thymosin, interferon, transfer factor, BCG vaccine polysaccharide, and any kind of bacterial extract such as Biostim, pneumonia vaccine, and influenza vaccine).
* Currently pregnant or breast-feeding women, or those who have fertility but cannot take contraceptive measures during the study period.
* Other conditions that are not suitable for the trials according to investigator's judgement.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
AECOPD (Acute exacerbation COPD) | 12 months
  Incidence of AECOPD within 12 months. Diagnosis of AECOPD is based on the Chinese Expert Consensus on Diagnosis and Management of AECOPD (2023 version).
  * Mild：No respiratory failure. Respiratory rate 20-30 times/min; no use of ventilator or change in mental state; fraction of inspiration O2 (FiO2) improves after supplemental oxygen; no increase in partial pressure of CO2 in artery (PaCO2).
  * Moderate：Acute respiratory failure but not life threatening. Respiratory rate > 30 times/min; use of ventilator or change in mental state; FiO2>35% after supplemental oxygen, improved hypoxemia; hypercapnia, PaCO2 increases from baseline or increases to 50-60mmHg.
  * Severe：Acute respiratory failure and life threatening. Respiratory rate > 30 times/min; use of ventilator; acute changes in mental state; FiO2>45% after supplemental oxygen, no improvement in hypoxemia; PaCO2 increases by > 60mmHg from baseline or acidosis.

SECONDARY OUTCOMES:
Moderate or severe AECOPD | 12 months
  Incidence of moderate or severe AECOPD within 12 months. Diagnosis of AECOPD is based on the Chinese Expert Consensus on Diagnosis and Management of AECOPD (2023 version).
Change in frequency of AECOPD | 12 months
  Change in frequency of AECOPD within 12 months. Diagnosis of AECOPD is based on the Chinese Expert Consensus on Diagnosis and Management of AECOPD (2023 version).
Hospitalization due to severe AECOPD | 12 months
  Hospitalization due to severe AECOPD within 12 months. Diagnosis of AECOPD is based on the Chinese Expert Consensus on Diagnosis and Management of AECOPD (2023 version). Hospitalization include ICU admission.
mMRC（modified Medical Research Council） | 1 month, 3 months, 6 months, and 12 months
  Changes in mMRC during the observation period. mMRC score a 5-point (0-4) scale, and higher grades indicate higher severity of dyspnea.
CAT（COPD Assessment Test） | 1 month, 3 months, 6 months, and 12 months
  Changes in CAT during the observation period. CAT score ranges from 0 to 40 points, and higher scores indicate higher symptom burden of COPD on patients.
TDI（Transition Dyspnea Index） | 1 month, 3 months, 6 months, and 12 months
  Changes in TDI during the observation period. TDI score ranges from -9 to 9 points, and higher scores indicate more significant improvements from baseline.
CET（Cough Evaluation Test） | 1 month, 3 months, 6 months, and 12 months
  Changes in CET during the observation period. CET score ranges from 5 to 25 points, and higher scores indicate higher cough severity.
Cough severity VAS（Visual Analog Scale） | 1 month, 3 months, 6 months, and 12 months
  Changes in VAS during the observation period. VAS a 100-mm linear scale ranging from "no cough" (0 mm) to "worst cough" (100 mm), and higher scores indicate higher cough severity.
Changes in the use of inhaled drugs | 1 month, 3 months, 6 months, and 12 months
  According to the medication administration record, any changes in the use of inhaled drugs during the observation period, including dosage, frequency, duration, etc.
Pulmonary function | 6 months, and 12 months
  Changes in pulmonary function during the observation period. Pulmonary function is evaluated by the ratio of forced expiratory volume in the first second (FEV1) to forced vital capacity (FVC) (FEV1/FVC)
Changes in the use of anti-infective drugs | 12 months
  According to the medication administration record, any changes in the use of ianti-infective drugs within 12 months, including dosage, frequency, duration, etc.
Adverse events | 12 months
  Occurrence of any Staphylococcus and Neisseria related adverse events during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang Sun, M.D., Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China